CLINICAL TRIAL: NCT02318628
Title: Advanced Approach to Arterial Stiffness (AAA Study - Triple A Study)
Brief Title: Advanced Approach to Arterial Stiffness
Acronym: AAA
Status: Completed | Type: Observational
Sponsor: International Society for Vascular Health (Other)
Responsible Party: Sponsor
Other Study IDs: ISVH3A2013
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Arterial Stiffness
Keywords: Cardio ankle vascular index; CAVI; pulse wave velocity; PWV; Non invasive arterial structure assessment
MeSH Terms: interventions — Cardio Ankle Vascular Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cardio Ankle Vascular Index (CAVI) of the Vasera system VS1500N — CAVI will be measured using the Vasera device (VS1500 n - Fukuda Denshi co, Japan). This device is easy to use and calculates automatically the CAVI.
  CAVI measurements will be performed according to the manufacturer Measurements will be performed after five to ten minute - period of rest in order to obtain a steady hemodynamic state and to limit measurements variability.

SUMMARY:
The aim of the 3A Study is to assess the role of MetS on the arterial mechanics and vascular health in different age groups using the Cardio Ankle Vascular Index (CAVI) of the Vasera system and the "classic" carotid-femoral Pulse Wave Velocity (PWV).

DETAILED DESCRIPTION:
Hypothesis The aim of thie 3A study is to assess the role of MetS on the arterial mechanics and vascular health in different age groups using the Cardio Ankle Vascular Index (CAVI) of the Vasera system and the "classic" carotid-femoral Pulse Wave Velocity (PWV).

STUDY OBJECTIVES

1. Objectives Primary Objective: Assess the influence of MetS on CAVI values (primary study endpoint) in 3 different age groups (40-54, 55-69, 70-85 years) of a European population.
2. Secondary Objectives

   * Establish the CAVI values in a European population according to the clusters of (MetS) components i.e. cardiovascular risk factors: abdominal obesity, high triglycerides, low HDL cholesterol, elevated blood pressure (BP), systolic or diastolic, and elevated fasting glucose (and diabetes), as well as tobacco smoking.
   * Assess the correlation between CAVI and the carotid-femoral PWV in the full population and in each age group; and compare the impact of MetS and its components on both the CAVI and PWV
   * To establish, the relationship between cardiovascular risk factors and the evolution of arterial stiffness as evaluated by CAVI and carotid-femoral PWV over a 2-year follow-up period.
   * To assess changes and predictive value of CAVI on organ damages and CV events during the follow-up period.
   * To assess 24h ABPM and its correlations and variations with the CAVI and PWV in patients with MetS and/or its different components.

This is a multinational European prospective longitudinal study.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 40-85 with life expectancy over 2 years will be included. Patients will be stratified according to their age (3 groups: 40-54, 55-69, 70-85 years)) and the presence or not of MetS.

Exclusion Criteria:

* Factors that may impair the quality of the CAVI and /or the PWV measurement or make PWV recording unreliable: known significant peripheral vascular disease with proximal artery stenosis, ankle brachial index < 0.9, or limb amputation; history of vascular surgery at the level of the carotid artery, femoral artery or aorta; body mass index > 40 kg/m²; atrial fibrillation and/or other major arrhythmia.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 40-85 with life expectancy over 2 years will be included. Patients will be stratified according to their age (3 groups: 40-54, 55-69, 70-85 years)) and the presence or not of MetS.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2014-12-01; Primary Completion 2016-06-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Cardio-Ankle-Vascular Index | 2 years
  CAVI will be measured using the Vasera device (Fukuda Denshi co, Japan). This device is easy to use and calculates automatically the CAVI.
  CAVI measurements will be performed according to the manufacturer recommendations Measurements will be performed after five to ten minute - period of rest in order to obtain a steady hemodynamic state and to limit measurements variability.
  The details of the CAVI measurements are shown in a specific document, C.F. appendix
  Ankle Brachial Index (ABI):
  The Ankle Brachial Index (ABI) will be measured using the Vasera device (Fukuda Denshi co, Japan). This device will calculate the ABI automatically.
  ABI measurements will be performed according to the manufacturer recommendations Measurements will be performed after five to ten minute - period of rest in order to obtain a steady hemodynamic state and to limit measurements variability.

SECONDARY OUTCOMES:
Pulse Wave Velocity | 2 years
  Measurement of PWV will be performed using a validated automatic device (Complior®, Sphygmocor®, and PulsePen®). The method of "simultaneous" recordings of the pulse waves from 2 different sites (carotid and femoral arteries) will be preferred. Because of the use of several devices, normalisation of the measurement values will be performed according to the European Experts recommendations.
Blood pressure Measurements | 2 YEARS
  Blood pressure will be measured in clinic according to the European Society of Hypertension (ESH) guidelines. BP should be measured in a standardized fashion using equipment that meets certification criteria.

CONTACTS AND LOCATIONS:
Overall Officials: JIRAR TOPOUCHIAN, Study Director — ISVH
Locations (1):
- ISVH, Paris, France